CLINICAL TRIAL: NCT05634499
Title: A Phase II, Single-Arm Study of Giredestrant in Patients With Grade 1 Endometrial Cancer
Brief Title: A Study of Giredestrant in Participants With Grade 1 Endometrial Cancer
Acronym: EndomERA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO44195; 2022-002443-21 (EudraCT Number); 2023-504091-23-00 (Other: EU Trial Number)
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — giredestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Giredestrant (Experimental)
  Interventions: Drug: Giredestrant

INTERVENTIONS:
Drug: Giredestrant — Participants will receive giredestrant 30 milligrams (mg) taken orally (PO) once a day (QD) on Days 1 to 28 of each 28-day cycle for 6 cycles. After completion of 6 cycles, the participant and investigator can choose to continue study treatment for an additional 18 cycles or discontinue study treatment and receive investigator-determined care.
  Other Names: RO7197597; GDC-9545; RG6171

SUMMARY:
This Phase II, global, single-arm study is designed to evaluate the efficacy, safety, and pharmacokinetics of giredestrant monotherapy in participants with Grade 1 endometrioid endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Grade 1 endometrial cancer (EC) of endometrioid histology for which participants are willing to receive 6-cycles of study therapy. An endometrial biopsy (EMB) or dilation and curettage (D&C) fresh collected within the screening period or archival sample collected within 3 months prior to screening must be provided to a central laboratory for histologic confirmation to determine eligibility.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Magnetic resonance imaging (MRI)-confirmation of non-deeply invasive tumor (<50% myometrial invasion)
* MRI or computed tomography (CT)-confirmation of no extrauterine disease
* Willing to undergo a minimum of 6 continuous cycles of therapy before decision on surgery
* No prior treatment for endometrial cancer
* Able and willing to take oral medications
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Adequate hematologic and end-organ function, as defined in the protocol
* Negative HIV test at screening, with the following exception: Patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥200/μL, and have an undetectable viral load.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agree to refrain from donating eggs, during the treatment period and for 30 days after the final dose of giredestrant, as defined in the protocol

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 30 days after the final dose of giredestrant or within the time period specified per local prescribing guidelines after the final dose of the investigator's choice of endocrine therapy
* Participants with non-endometrioid histologies, such as serous, clear cell, and mixed
* Treatment with investigational therapy within 28 days prior to initiation of study enrollment
* Treatment for cancer including but not limited to, chemotherapy, immunotherapy, cyclin-dependent kinase (CDK)4/6 inhibitors, endocrine therapy, biologic therapy, or herbal therapy within 28 days prior to the initiation of study enrollment
* Any gastrointestinal condition causing malabsorption or obstruction (e.g., celiac sprue, gastric bypass surgery, strictures, adhesions, history of small bowel resection, blind loop syndrome)
* Known hypersensitivity to giredestrant or its excipients
* Known intercurrent illness or psychiatric illness/social situations that will limit compliance with study requirements
* Evidence or high suspicion of metastatic/extrauterine disease at enrollment
* Unwilling or unable to comply with study-related procedures, including all endometrial sampling/biopsies
* Planned surgery, either for the treatment of cancer or any other surgery, during the study treatment period and up to 10 days after the completion of study treatment
* Serious infections requiring IV antibiotics within 7 days prior to initiation of study treatment or any active infection that, in the opinion of the investigator, could impact participant safety
* Participants who have clinically significant liver disease consistent with Child-Pugh Class B or C, including active hepatitis (e.g., hepatitis B virus [HBV] or hepatitis C virus [HCV]), current alcohol abuse, cirrhosis, or positive test for viral hepatitis, as defined in the protocol
* Treatment with strong CYP3A4 inhibitors or inducers within 14 days or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment
* Any serious medical condition or abnormality in clinical laboratory tests that precludes the participant's safe participation in and completion of the study
* History of other malignancy within 5 years prior to screening, except for those with an expected negligible risk for metastases or death (e.g., 5-year overall survival 90%) after curative treatment
* Active tuberculosis
* Severe infection per investigator judgment at the time of enrollment, including but not limited to, use of systemic antibiotics, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion of the investigator, could impact participant safety
* Significant cardiovascular disease, such as cardiac disease New York Heart Association Class II or greater, myocardial infarction, or cerebrovascular accident within 3 months prior to enrollment, unstable arrhythmias, or unstable angina
* Active cardiac disease or history of cardiac dysfunction, as defined in the protocol
* Major surgical procedure other than for diagnosis within 28 days prior to enrollment or anticipation of need for a major surgical procedure during the study
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the participant at high risk for treatment complications illnesses or conditions that interfere with the participant's capacity to understand, follow, and/or comply with study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Have Regression at 6 Months | Baseline, 6 Months
  The percentage of participants who have regression is defined as participants who have a decrease in the proportion of cancer in their endometrial biopsy or the proportion of cancer is not increased, but there is an increase in non-cancer/non-atypical hyperplasia at the 6-month assessment compared with baseline.
Number of Participants with at Least One Adverse Event, with Severity Determined According to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0) | From Baseline until 30 days after the final dose of study drug (up to 1 year, 6 months)

SECONDARY OUTCOMES:
Percentage of Participants Who Have Complete Regression at 6 Months | Baseline, 6 Months
  The percentage of participants who have complete regression is defined as participants having an assessment of 100% of non-cancer/non-atypical hyperplasia at the Month 6 assessment.
Median Duration of Regression | From first regression to first relapse (up to 1 year, 6 months)
Median Time to First Regression | From first study treatment to first regression (up to 1 year, 6 months)
Median Time to Relapse or Loss of Clinical Benefit | From first study treatment to relapse or loss of clinical benefit, whichever occurs first (up to 1 year, 6 months)
Plasma Concentration of Giredestrant at Specified Timepoints | Predose on Day 1 of Cycles 1, 2, 3, 4, and 6; 3-4 hours Postdose on Day 1 of Cycles 1 and 2 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (7):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Minnesota Oncology Minneapolis, Minneapolis, Minnesota
  - Englewood Health/Hematology Oncology Practice of Englewood (HOPE), Englewood, New Jersey
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST - PPDS, Meldola, Emilia-Romagna, Italy
- Poland (2):
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice, Gliwice
  - Swietokrzyskie Centrum Onkologii, Kielce

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing